CLINICAL TRIAL: NCT01639625
Title: Open Clinical Trial, Uncontrolled in Patients Bearing Squamous Cell Carcinoma or Adenocarcinoma of the Cervix Stage IIA and IIB FIGO Classification Treated With Radiotherapy External Endocavitary Brachytherapy + Concurrent Hemotherapy Weekly Systemic and Local Application of CIGB-300 Dose Escalation
Brief Title: Concurrent Treatment of Squamous Cell Carcinoma or Adenocarcinoma of the Cervix With CIGB-300 for Local Application
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laboratorio Elea Phoenix S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 300CX02AR01
Record Dates: First submitted 2012-06-15; First posted 2012-07-13 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-08

CONDITIONS: Squamous Cell Carcinoma of the Cervix; Adenocarcinoma of the Cervix
MeSH Terms: interventions — CIGB-300

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CIGB300 (Experimental)
  Interventions: Drug: CIGB300

INTERVENTIONS:
Drug: CIGB300 — CIGB300: 15 mg, 35 mg and 70 mg All groups will receive CIGB-300 for local application.

SUMMARY:
They include patients who are candidates to complete concurrent treatment with endocavitary brachytherapy External radiation therapy + more QT based weekly cisplatin.

ELIGIBILITY:
Inclusion Criteria:

* Stages IIA and IIB FIGO classification.
* Age between 21 to 70 years.
* ECOG performance status 0-1.
* No history of another neoplastic disease.
* Value of Hemoglobin ≥ 9 g / l.
* Total leukocyte count ≥ 3.0 x 109 / L.
* Absolute neutrophil count ≥ 1.5 x 109 / L.
* Platelets ≥ 100,000 x mm3.
* Total bilirubin ≤ 1.5 times ULN, SGOT and SGPT ≤ 2.5 times upper limit of normal.
* Creatinine ≤ 2 mg / dL and creatinine clearance calculated ≥ 60 ml / min(according to Cockcroft-Gault formula)
* Patients of childbearing age who are using an adequate contraception method during treatment to prevent pregnancy.
* Life expectancy ≥ 12 months
* Measurable disease
* Informed consent signed by the patient

Exclusion Criteria:

* Pregnancy and lactation period.
* Presence of lymph node metastases or hematogenous extrapelvic known.
* Uncontrolled intercurrent diseases, including active infection, symptomatic congestive heart failure, unstable angina or cardiac arrhythmia and psychiatric illness involving incompetence of the patient.
* Other malignancies, with the exception of basal cell carcinoma or other tumor that appropriate treatment is received showing a disease-free period ≥ 5 years.
* Hepatitis B or C active, positive serology for HIV.
* Atopy history of severe / severe asthma.
* A history of autoimmune disease.
* Presence of significant abnormalities in ECG performed within 14 days prior to admission.
* Diseases that prevent the patient give informed consent or their ability to collaborate in the trial.
* Participating in another clinical trial "

Ages: 21 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-05; Primary Completion 2015-09 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with presence or absence of grade 3 or 4 adverse events related to the study drug, in each dose level | Up to 2 years

SECONDARY OUTCOMES:
Number of patients with local relapses | Up to 2 years
Number of patients with distant relapses | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Oncologia Angel H. Roffo, Ciudad Autonoma de Buenos Aires, Buenos Aires, Argentina